CLINICAL TRIAL: NCT03016260
Title: Proof-of-Performance Study of RABIOPRED Assay as an In Vitro Diagnostic Test to Identify Patients With Rheumatoid Arthritis Who Are Unlikely to Show Response to 1st Treatment With Anti-TNFα and Methotrexate Combination.
Brief Title: RABIOPRED - a Validation Study of Theranostic Test to PREDict Treatment Response of Anti-TNFα BIologicals in Rheumatoid Arthritis
Acronym: RABIOPRED
Status: Terminated | Type: Observational
Sponsor: TcLand Expression S.A. (Industry)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-A00556-45
Record Dates: First submitted 2017-01-04; First posted 2017-01-10 (Estimated); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: RheumatoId Arthritis
Keywords: Rheumatoid Arthritis; Anti TNF; Infliximab; Adalimumab; Etanercept; Golimumab; Certolizumab Pegol; Infliximab biosimilar; Etanercept biosimilar; Methotrexate
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab; Adalimumab; Etanercept; golimumab; Certolizumab Pegol; CT-P13; etanercept biosimilar SB4

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA, RNA, Plasma, Serum, PBMC and Urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (8):
- Infliximab (Remicade®)
  Interventions: Biological: Infliximab
- Adalimumab (Humira®)
  Interventions: Biological: Adalimumab
- Etanercept (Enbrel®)
  Interventions: Biological: Etanercept
- Golimumab (Simponi®)
  Interventions: Biological: Golimumab
- Certolizumab Pegol (Cimzia®)
  Interventions: Biological: Certolizumab Pegol
- Infliximab biosimilar (Remsima®/ Inflectra®)
  Interventions: Biological: Infliximab biosimilar
- Etanercept biosimilar (Benepali®)
  Interventions: Biological: Etanercept biosimilar
- Infliximab biosimilar (Flixabi®)
  Interventions: Biological: Infliximab biosimilar

INTERVENTIONS:
Biological: Infliximab — Anti-TNF alpha originator
  Other Names: Remicade®
  Groups: Infliximab (Remicade®)
Biological: Adalimumab — Anti-TNF alpha originator
  Other Names: Humira®
  Groups: Adalimumab (Humira®)
Biological: Etanercept — Anti-TNF alpha originator
  Other Names: Enbrel®
  Groups: Etanercept (Enbrel®)
Biological: Golimumab — Anti-TNF alpha originator
  Other Names: Simponi®
  Groups: Golimumab (Simponi®)
Biological: Certolizumab Pegol — Anti-TNF alpha originator
  Other Names: Cimzia®
  Groups: Certolizumab Pegol (Cimzia®)
Biological: Infliximab biosimilar — Anti-TNF alpha Infliximab biosimilars
  Other Names: Remsima® or Inflectra®
  Groups: Infliximab biosimilar (Remsima®/ Inflectra®)
Biological: Etanercept biosimilar — Anti-TNF alpha Etanercept biosimilar
  Other Names: Benepali®
  Groups: Etanercept biosimilar (Benepali®)
Biological: Infliximab biosimilar — Anti-TNF alpha Infliximab biosimilar
  Other Names: Flixabi®
  Groups: Infliximab biosimilar (Flixabi®)

SUMMARY:
RABIOPRED is an in vitro non-invasive blood test, which aims to identify patients with rheumatoid arthritis (RA) who are not likely to respond to anti-TNFα and methotrexate combination therapy.

DETAILED DESCRIPTION:
Multi-centre, non-interventional, open-label, non-comparative, prospective cohort study with a clinical follow-up between (a) 12 and 14 weeks and (b) 22 and 24 weeks.

The RABIOPRED test is indicated for use in patients:

* 18 years of age or older,
* Eligible for a first line biologic therapy with anti-TNF alpha. The RABIOPRED test is indicated for use by rheumatologists as a biological basis for guiding anti-TNF alpha treatment prior to its initiation.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a confirmed Rheumatoid Arthritis according the American College of Rheumatology (ACR) classification criteria (Arnett FC, 1988, Arthritis Rheum)
* Patient with a DAS28 index greater than 3.2.
* Patient eligible for treatment with an anti-TNFα agent (any one of Remicade®, Humira®, Enbrel®, Simponi®, Cimzia®, Remsima®/Inflectra®, Benepali® and Flixabi® according to the "Summary of Product Characteristics" for each product) and Methotrexate combination therapy,
* Patient refractory to treatment with at least one classical DMARDs (one of which has to be MTX) prescribed according to the international recommendations, i.e. for at least 12 weeks at the maximal tolerated dose prior to anti-TNFα treatment and with doses which must have been kept stable during the 4 weeks preceding the initiation of the anti-TNFα therapy. In case of Leflunomide treatment, patients may be included in the study after a period of at least 3 months of Leflunomide stop, or after a washout by cholestyramine for at least 11 days.
* Use of oral steroids (≤ 10 mg/day of prednisone or equivalent dose of another molecule) and/or NSAIDs will be permitted; doses must have been kept stable during the 4 weeks preceding the initiation of the anti-TNFα therapy
* Patient (male or female) at 18 years of age or older at inclusion,
* Negative β-HCG (Human Chorionic Gonadotrophin) pregnancy test, when appropriate, according to the patient's age and contraceptive method.
* Written Informed consent signed from the patient.

Exclusion Criteria:

* Patient having received previously any anti-TNFα biologic therapy or any molecule in development belonging to anti-TNFα class. Patients having received other biologics (such as anti-CD20, anti-CTLA4, IL1 blockers, IL6 blockers and other molecules in development) can be included in the study after a period of at least 6 months,
* Patient non eligible to anti-TNFα according to the SmPC (Summary of Products),
* Patient on anti-TNFα monotherapy without methotrexate,
* Patient with clinically significant, severe and uncontrolled infectious diseases,
* Patient with symptoms of a significant somatic or psychiatric/mental illness,
* Patient with other auto-immune diseases (i.e. Inflammatory Bowel Diseases, Systemic Lupus Erythematosus, vasculitis, uncontrolled asthma, etc.),
* Patient with evidence of cardiac, pulmonary, metabolic, renal, hepatic, gastro-intestinal conditions, which, in the opinion of the Investigator, may interfere with the study,
* Cancer,
* Pregnancy,
* Nursing mothers,
* Patient who is participating in a clinical trial of other biologics or for whom a period of exclusion has been defined

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from rheumatoid arthritis eligible for biologic therapy, for whom the rheumatologist envisages anyone of anti-TNFα, will be included in this study. As the study should not modify patient care, it is not authorized to prescribe study biologics if other biologic is considered for a given patient or if a given patient is not eligible for study biologic treatment.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
EULAR response criteria | 13th week (+/- 7 days)
  Performance of RABIOPRED test to predict treatment response of anti-TNFα agents based on the EULAR (EUropean League Against Rheumatism) response criteria at 13th week (+/- 7 days) compared with baseline.

SECONDARY OUTCOMES:
ACR response criteria | 13th week (+/- 7 days)
  Performance of RABIOPRED test to predict treatment response of anti-TNFα agents based on ACR (American College of Rheumatology) response criteria at 13th week (+/- 7 days) compared with baseline.
EULAR response criteria | 23rd week (+/- 7 days) or at the time of treatment switch
  Performance of RABIOPRED test to predict treatment response of anti-TNFα agents based on the EULAR (EUropean League Against Rheumatism) response criteria at 23rd week (+/- 7 days) or at the time of treatment switch (whichever comes first) compared with baseline.
SDAI (Simplified Disease Activity Index) score | 23rd week (+/- 7 days) or at the time of treatment switch
  Performance of RABIOPRED test to predict treatment response of anti-TNFα agents based on achieving Low Disease Activity (LDA) according to SDAI score at 23rd week (+/- 7 days) or at the time of treatment switch (whichever comes first) compared with baseline.

CONTACTS AND LOCATIONS:
Locations (8):
- Institute of Rheumatology, Prague, Czechia
- France (3):
  - CHU-Montpellier, Montpellier
  - CHU Nice, Nice
  - CHU Strasbourg Hautepierre, Strasbourg
- Tel Aviv Surasky Medical Center, Tel Aviv, Israel
- Leiden University Medical Center, Leiden, Netherlands
- Turkey (Türkiye) (2):
  - Istanbul University, Istanbul
  - University of Marmara, Istanbul